CLINICAL TRIAL: NCT06052813
Title: A PhaseI/II, Multicenter, Open-label Clinical Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of the Menin Inhibitor BN104 in the Treatment of Patients With Relapsed/Refractory Acute Leukemia
Brief Title: A Study of BN104 in the Treatment of Acute Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BN104-101
Record Dates: First submitted 2023-09-06; First posted 2023-09-25 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: ALL, Adult; AML, Adult; Acute Leukaemia; KMT2A Rearrangement; NPM1 Mutation; NUP98 Gene Rearrangement; Menin Inhibitors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- 200mg QD (Experimental): The starting dose cohort(200mg QD) where accelerated titrated dose-escalation method is applied, a patient will initially receive a single dose BN104 on Day 1 of Cycle 0 (3 days prior to Day 1 of Cycle 1) to evaluate the concentration of BN104 up to 72 hours after administration and the safety of single dose of BN104. Then the patient begins continuous treatment with BN104 200 mg QD on Day 1 of Cycle 1 by every 28-day treatment cycle until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- 200mg BID (Experimental): After completion of DLT evaluation for the first dose cohort (200 mg QD), patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- 400mg BID (Experimental): After completion of DLT evaluation for the first dose cohort (200 mg QD), patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- 600 BID (Experimental): After completion of DLT evaluation for the first dose cohort (200 mg QD), patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- 800 BID (Experimental): After completion of DLT evaluation for the first dose cohort (200 mg QD), patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- Adolescent cohort - 400mg BID (Experimental): The first 3-6 patients will be dosed at 400 mg BID. If there is no significant difference in Cmax and AUC between adolescent and adult patients, and no DLT occurs in 3-6 patients or ≤1 DLT occurs in 6 patients, the dose will be escalated to 600 mg BID, and 3-6 additional adolescent patients will be enrolled. patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first.
  Interventions: Drug: BN104 monotherapy
- Adolescent cohort - 600mg BID (Experimental): patients will begin to receive twice daily (BID) dosing frequency in each 28-day treatment cycle for the subsequent dose cohorts for which conventional 3+3 design is used until disease progression, intolerable toxicity, withdrawal of consent, loss to follow-up, death, or other conditions in which patients are not suitable for study treatment, whichever occurs first. If ≤1 DLT occurs in 6 patients, at 600mg bid, then enrolment will be expanded at the 600 mg BID dose level to approximately 20 patients, for patients with relapsed/refractory acute leukaemia with KMT2A rearrangement and NPM1 mutation, ensuring at least 10 patients each with KMT2A rearrangement and NPM1 mutation in relapsed/refractory acute leukaemia at the 600 mg BID dose level.
  Interventions: Drug: BN104 monotherapy
- Phase II CohortA - Patients with relapsed/refractory AML with NPM1 mutation (Experimental): receiving oral BN104 treatment at a dose of 600 mg BID (300 mg BID when co-administered with strong CYP3A4 inhibitors)
  Interventions: Drug: BN104 monotherapy - rp2d
- Phase II Cohort B: r/r acute leukaemia with KMT2Ar (including AML, ALL, or MPL) (Experimental): receiving oral BN104 treatment at a dose of 600 mg BID (300 mg BID when co-administered with strong CYP3A4 inhibitors)
  Interventions: Drug: BN104 monotherapy - rp2d

INTERVENTIONS:
Drug: BN104 monotherapy — Phase I(adults): Will be administered orally once daily (approximately every 24 hours) for the first cohort or twice daily (approximately every 12 hours) for the subsequent cohorts.
  Arms: 200mg BID; 200mg QD; 400mg BID; 600 BID; 800 BID
Drug: BN104 monotherapy — Phase I(adolescent): Will be administered orally twice daily (approximately every 12 hours)
  Arms: Adolescent cohort - 400mg BID; Adolescent cohort - 600mg BID
Drug: BN104 monotherapy - rp2d — receiving oral BN104 treatment at a dose of 600 mg BID (300 mg BID when co-administered with strong CYP3A4 inhibitors)
  Arms: Phase II Cohort B: r/r acute leukaemia with KMT2Ar (including AML, ALL, or MPL); Phase II CohortA - Patients with relapsed/refractory AML with NPM1 mutation

SUMMARY:
The Phase I/II trial is to learn the safety, pharmacokinetics, and preliminary efficacy of BN104 taken once daily or twice daily in patients with acute lymphocytic leukemia or acute myeloblastic leukemia.

DETAILED DESCRIPTION:
The study is divided into 2 phases. Phase1 part will enroll 98 patients to evaluate safety and tolerance of BN104 in patients with relapsed/refractory (R/R) Acute Leukemia to determine maximum tolerated dose and recommended phase2 dose (RP2D), including approximately 66 adult patients and 32 adolescent patients with specific mutations (KMT2A gene rearrangement, NPM1 gene mutation, NUP98 mutation) enrolled at phaseI.

Phase II expansion part will enroll 168 patients and be conducted at the selected dose level to further evaluate the safety and tolerability of BN104, as well as preliminary efficacy in Acute leukemia subjects with specific mutations (KMT2A gene rearrangement or NPM1 gene mutation). Patients will be allocated into 2 Acute Leukemia subgroup cohorts depends on their genotype.

* Cohort A: Patients with Relapsed/refractory AML subjects with NPM1 mutations
* Cohort B: Patients with relapsed/refractory acute leukaemia with KMT2A rearrangement (including AML, ALL, or MPL)

Patients will receive orally administrated BN104 once daily or twice daily. Study drug will be administered in 28-day cycles until disease progression or unacceptable toxicity, death, Informed consent withdraw ect.

Laboratory tests will be performed weekly in Cycles 1-2, bi-weekly in Cycle3 and every 4weeks from Cycle 4 onwards. Efficacy assessment will be performed on baseline, C2D1, C3D1 and every 2 cycles from Cycle3 onwards. Additional clinical assessments and laboratory tests may be performed at discretion of the investigator as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Have been fully informed about the study and have voluntarily signed the ICF;
2. Patients diagnosed with relapsed/refractory acute leukaemia (including AML, ALL, and mixed-phenotype acute leukaemia, excluding acute promyelocytic leukaemia) according to the World Health Organization (WHO) criteria in 2022, with bone marrow morphological changes (blasts/immature cells ≥ 5%), and who have been evaluated by the investigator to have no better treatment options, must meet at least one of the following conditions:

   * Primary refractory disease, newly diagnosed disease that show no response after 2 cycles of standard treatment;
   * First relapse, relapsed within 12 months after CR/CRh/CRi following consolidation/intensive therapy;
   * Relapsed after 12 months and unresponsive to conventional salvage chemotherapy;
   * Patients with 2 or more relapses;
   * Patients intolerant to intensive chemotherapy who experience disease progression during continuous low-intensity therapy; Note: Patients with secondary AML or AML transformed from MDS, MPN, can also be enrolled, but they need to meet the above criteria after the disease has transformed into AML;
3. For all Phase I patients, the presence of NPM1 mutation, or KMT2A rearrangement, or NUP98 rearrangement must be confirmed,During Phase I, patients with other acute leukemia subtypes shown to depend on menin-KMT2A interaction (e.g., UBTF-TD) or driven by HOXA/MEIS1 overexpression may also be eligible after consultation with the Sponsor's Medical Monitor;
4. Patients in the Phase II (single-arm pivotal clinical study) must have a confirmed NPM1 mutation or KMT2A rearrangement. Enrollment based on local testing results is acceptable with a copy of the test report provided; however, all patients are required to submit screening bone marrow samples to the central laboratory ,Eligible NPM1 mutations include exon12 type A, B, and D mutations ; other NPM1 mutations causing cytoplasmic localization require sponsor pre-approval for enrollment. KMT2A rearrangements exclude non-fusion rearrangements involving KMT2A partial tandem duplication (KMT2A-PTD).
5. Peripheral blood white blood cell count ≤ 35 × 109/L (use of hydroxyurea to control peripheral white blood cell count is permitted);
6. Age ≥ 12 years (for adolescent patients aged 12 years or older but not yet 18 years old, weight must be ≥ 40 kg);
7. ECOG score 0-2;
8. Adequate hepatic, renal, and cardiac functions
9. Expected survival of more than 12 weeks as judged by the investigator
10. For patients with D-dimer test results > 5 × ULN during screening, relevant tests (such as rechecking coagulation function after a certain interval, lower extremity deep vein ultrasound, etc.) are required to exclude deep vein thrombosis, hypercoagulation, and disseminated intravascular coagulation before enrollment;
11. Able to undergo treatment, visits, and study-related examinations as required by the protocol;
12. Female patients of childbearing potential or male patients whose female partners are of childbearing potential must agree to use effective methods of contraception during the study and for 30 days after the last dose of study drug, such as double barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. Postmenopausal women (> 45 years old and amenorrheic for more than 1 year) and surgically sterilized women are not subject to this condition.

Exclusion Criteria:

1. Known active central nervous system (CNS) leukaemia (including imaging abnormalities and CSF smear or flow cytometry indicating leukaemia cells; prior CNS leukaemia that has been treated and controlled is acceptable, but requires screening lumbar puncture and CSF test for confirmation, or routine standard CNS prophylaxis is acceptable);
2. Known history of clinically significant liver disease, including viral or other hepatitis or hepatic cirrhosis:

   * Hepatitis B surface antigen (HBsAg) seropositive, requires Hepatitis B virus (HBV) DNA negative for enrollment;
   * For Hepatitis C virus (HCV) antibody seropositive patients, HCV RNA negative result is required for enrollment.
3. Known human immunodeficiency virus (HIV) infection;
4. Pregnancy (positive pregnancy test at screening) or lactating females;
5. Any of the following cardiac-related criteria is met:

   * Hereditary long QT syndrome or QTcF > 450 msec;
   * Various clinically significant cardiovascular disorders, including acute myocardial infarction, unstable angina pectoris, coronary artery bypass surgery within 6 months prior to enrollment, cardiac failure congestive of New York Heart Association (NYHA) Class 2 or higher (including Class 2), etc.;
6. Patient has other concomitant malignant tumours, except for:

   * Curatively treated skin basal cell carcinoma, breast cancer in situ, or cervical carcinoma in situ, etc.;
   * Patients with low-grade lymphoma who are in CR, asymptomatic, without large mass lesions, and do not require systemic therapy or radiotherapy;
   * Other malignant tumours treated with curative intent, with CR achieved for at least 2 years, and no requirement for systemic maintenance therapy or radiotherapy;
7. Received autologous haematopoietic stem cell transplant (ASCT) or Chimeric Antigen Receptor T-cell (CAR-T) therapy within 60 days prior to screening, or toxicity related to ASCT or CAR-T therapy has not yet resolved;
8. Underwent allogeneic HSCT within 100 days prior to screening, or the patient still has Grade ≥ 2 acute graft versus host disease or chronic graft versus host disease requiring systemic treatment, or the patient still requires immunosuppression (prednisone ≤ 10 mg/day or equivalent dose of other corticosteroids is permissible for screening; corticosteroids need to be gradually tapered and discontinued after enrolment unless there is a specific reason);
9. Received donor lymphocyte infusion (DLI) within 28 days prior to screening;
10. Prior anti-leukaemia therapy, including chemotherapy, radiotherapy, hormone therapy, targeted therapy, or immunotherapy (excluding hydroxyurea), etc., less than 2 weeks or 5 half-lives (whichever is shorter) before the start of study treatment;
11. Previous participation in other drug clinical studies, with less than 2 weeks or 5 half-lives since the last use of a small molecule drug, or less than 4 weeks or 5 half-lives for large molecule drugs (such as antibody drugs), whichever is shorter;
12. Previous treatment targeting menin;
13. Toxicity from previous anti-leukaemia therapy has not recovered to Grade 0 or 1 (except for alopecia and cytopenias reasonably considered related to the underlying disease);
14. Patients who had a chest CT scan within 1 month prior to screening showing pulmonary nodules need to undergo a T-SPOT.TB test (Tuberculosis infection T-cell spot test) during screening; those with a positive result must be excluded (no additional test required if no chest CT scan was performed within 1 month prior to screening);
15. Uncontrolled active infection:

    * Patients with non-severe infectious complications (such as oral candida infection or uncomplicated urinary tract infection) currently receiving oral/topical anti-infective therapy may be enrolled;
    * Patients with severe infection requiring hospitalisation or intravenous antibiotic therapy within 14 days prior to enrollment, patients with no evidence of infection receiving prophylactic anti-infective, anti-fungal, or anti-viral therapy due to prolonged neutropenia may be enrolled;
    * Patients receiving intravenous antibiotic therapy or hospitalized for febrile neutropenia, but with no evidence of infectious etiology found, and whose body temperature has been normal for more than 72 hours without antipyretics, may be enrolled;
16. Patient has known dysphagia, short-bowel syndrome, gastroparesis, or other conditions limiting oral drug intake or gastrointestinal absorption;
17. History of severe allergy to menin inhibitors or allergy to any component of BN104;
18. Investigator-judged insufficient compliance of the patient to participate in this clinical study;
19. Any other disease, metabolic abnormality, physical examination abnormal, or clinically significant laboratory test abnormal that, in the investigator's judgment, gives reason to suspect that the patient has a disease or condition unsuitable for the use of the study drug, or that will affect the interpretation of the study results, or place the patient at high risk.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PhaseI Incidence of Dose Dose limiting toxicities(DLTs) | DLT last 28days(at the end of cycle 1 for each dose)
  DLTs will be evaluated at the end of cycle 1(28 days after receiving BN104) for each dose level by evaluating abnormal laboratory examinations by the Investigator.
PhaseI Incidence of serious adverse events(SAEs) | 36 month
  SAEs will be recorded in the eCRF from time of the signing informed consent through 30 days after the last dose of BN104.
PhaseII efficacy assessment | 36 month
  To evaluate the efficacy of BN104 in treating patients with relapsed/refractory acute leukaemia with specific mutations (KMT2A rearrangement or NPM1 mutation) by mesuring patients bone marrow blasts/immature cells(CR, CRh rate) at protocol defined efficacy assessment timepoint

SECONDARY OUTCOMES:
Phase I/II Evaluate the number and frequency of adverse events (AEs) | 36 months
  Evaluate the number and frequency of adverse events (AEs) by evaluating abnormal laboratory examinations by the Investigator at each clinical visit from time of the signing informed consent through 30 days after the last dose of BN104.
Phase I/II Evaluate patient vital signs | 36 months
  Evaluate vital signs, including body temperature, heart rate, respiration rate, and blood pressure by the Investigator at each clinical visit before taking BN104.
Phase I/II Evaluate electrocardiogram (ECG) assessments | 36 months
  Evaluate electrocardiogram (ECG) assessments by the Investigator Prior to any examination at each clinical visit to monitor heart rate, R-R interval, QT interval and QTcF interval, QRS, and P-R interval times.
Phase I/II pharmacokinetic Maximum concentration (Cmax) | 36 months
  To characterized Maximum Plasma Concentration [Cmax] of BN104 by collecting and evaluating the serum at the protocol specified time points.
Phase I/II pharmacokinetic Peak time(Tmax) | 36 months
  To characterized Peak time(Tmax) of BN104 by collecting and evaluating the serum at the protocol specified time points
Phase I/II pharmacokinetic Clearance half-life (T1/2) | 36 months
  To characterized Clearance half-life (T1/2) of BN104 by collecting and evaluating the serum at the protocol specified time points
Phase I/II pharmacokinetic Area under the blood concentration-time curve (AUC0-t) | 36 months
  To characterized Area under the blood concentration-time curve (AUC0-t) of BN104 by collecting and evaluating the serum at the protocol specified time points.
Phase I/II pharmacokinetic metabolite M1 | 36 months
  To characterized BN104 major metabolite M1 by collecting and evaluating the serum at the protocol specified time points.
Phase I/II efficacy assessment based on Complete response (CR) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Complete response (CR) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based on Complete response with partial recovery of hematology (CRh) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Complete response with partial recovery of hematology (CRh) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based on Complete response with incomplete hematological recovery (CRi) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Complete response with incomplete hematological recovery (CRi) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment Objective response rate (ORR) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Objective response rate (ORR) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based on Duration of response (DOR) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Duration of response (DOR) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based on Event-free survival (EFS) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Event-free survival (EFS) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based Relapse-free survival (RFS) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based Relapse-free survival (RFS) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment based on Overall survival (OS) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Overall survival (OS) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
Phase I/II efficacy assessment Cumulative relapse rate (CIR) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Cumulative relapse rate (CIR) assessed by the Investigator at Cycle2. cycle3 and every 2 cycles thereafter through peripheral blood tests, detection of bone marrow primitive cell ratio and other morphological changes by bone marrow aspiration/biopsy
PhaseI pharmacokinetic biomarkers | 36 months
  Changes in pharmacokinetic biomarkers (e.g., HOXA9, MEIS1, CD11b, etc.) before and after BN104 administration, and correlations with dosing and efficacy
correlation between specific gene alterations and clinical efficacy | 36 months
  The correlation between specific gene alterations (such as NPM1 mutation, KMT2A rearrangement) and other gene alterations (such as FLT3 mutation/fusion, TP53 mutation, NUP98 fusion, etc.), and clinical efficacy.
Phase I/II efficacy assessment Cumulative Incidence of Death (CID) | 36 months
  To assess the preliminary anti-tumor activity of BN104 based on Cumulative Incidence of Death (CID) through the time from the date of achieving remission to non-relapse death

CONTACTS AND LOCATIONS:
Overall Officials: Depei WU, Prof., Principal Investigator — The First Affiliated Hospital of Soochow University; Mingyuan Sun, Dr., Principal Investigator — Institute of Hematology, Chinese Academy of Medical Sciences; Yan Li, Dr., Principal Investigator — Institute of Hematology, Chinese Academy of Medical Sciences; Xudong Wei, Prof., Principal Investigator — Henan Oncology Hospital; Dengju Li, Prof., Principal Investigator — Tongji Hospital; Yuhua Li, Prof., Principal Investigator — Southern Medical University, China; Xiaoyu Zhu, Prof., Principal Investigator — Anhui Provinvcal Hospital; Fei Li, Prof., Principal Investigator — The First Affiliated Hospital of Nanchang University; Jinhai Ren, Prof., Principal Investigator — The Second Hospital of Hebei Medical University; He Huang, Prof., Principal Investigator — Zhejiang University; Pengcheng He, Prof., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Wei Wang, Dr., Principal Investigator — The Affiliated Hospital of Qingdao University; Yu Cao, Dr., Principal Investigator — The Affiliated Hospital of Qingdao University; Songfu Jiang, Prof., Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Jian Ge, Prof., Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Bei Liu, Dr., Principal Investigator — LanZhou University; Yuping Gong, Prof., Principal Investigator — West China Hospital; Xiaojun Xu, Prof., Principal Investigator — Children's Hospital, Zhejiang University School of Medicine; Xiaofan Zhu, Prof., Principal Investigator — Chinese Academy of Medical Sciences Haematological Diseases Hospital; Wenting Hu, Dr., Principal Investigator — Shanghai Children's Medical Center; Meng LV, Dr., Principal Investigator — Peking University People's Hospital; Jun Luo, Prof., Principal Investigator — First Affiliated Hospital of Guangxi Medical University; Zhenfang Liu, Prof., Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No